CLINICAL TRIAL: NCT03168763
Title: Advanced Cancer Patients' Perception of Physician Compassion and Professionalism - A Randomized, Double Blind, Cross Over Trial
Brief Title: Effect of Physician Attire on Patients' Preference of Physician
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-0970; NCI-2018-01195 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Malignant neoplasms of independent (primary) multiple sites; Advanced Cancer; Videos; Questionnaires; Surveys
MeSH Terms: interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video 1A (Experimental): Questionnaires completed at baseline, after each video viewing, and at completion.
  Participants shown Video 1A or 1B, then shown Video 2A or 2B.
  Interventions: Behavioral: Video; Behavioral: Questionnaires
- Video 1B (Experimental): Questionnaires completed at baseline, after each video viewing, and at completion.
  Participants shown Video 1A or 1B, then shown Video 2A or 2B.
  Interventions: Behavioral: Video; Behavioral: Questionnaires
- Video 2A (Experimental): Questionnaires completed at baseline, after each video viewing, and at completion.
  Participants shown Video 1A or 1B, then shown Video 2A or 2B.
  Interventions: Behavioral: Video; Behavioral: Questionnaires
- Video 2B (Experimental): Questionnaires completed at baseline, after each video viewing, and at completion.
  Participants shown Video 1A or 1B, then shown Video 2A or 2B.
  Interventions: Behavioral: Video; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Video — Participants shown Video 1A or 1B, then shown Video 2A or 2B.
Behavioral: Questionnaires — Questionnaires completed at baseline, after each video viewing, and at completion.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn about the effects of a doctor's characteristics on participant's preference for a doctor. Researchers also want to learn about how a doctor's characteristics affect participant's options about professionalism and compassion.

DETAILED DESCRIPTION:
If participant agrees to take part in this study, participant will be asked to complete 7 questionnaires. These questionnaires ask about participant's gender, date of birth, ethnicity, marital status, level of education, religion, and information about the disease and treatments participant received. Participant will also be asked about any symptoms participant may be having, how much trust participant has in the medical profession in general, how participant feels about the disease, any depression or anxiety participant may have, and participant's level of hopefulness. These questionnaires should take about 6 minutes to complete.

Participant will be shown 2 videos (each 3 minutes long) and then participant will complete questions about each video. Participant will be asked to rate the doctors participant saw on their professionalism and their compassion.

Caregivers will be required to leave the room or stay silent while the participant is watching the videos.

The total time to watch the videos and complete the second set of questionnaires should be about 7 minutes.

Finally, participant will be asked to complete 3 questionnaires about participant's overall preference for a doctor. These questionnaires will take about 5 minutes to complete.

Length of Study Participation:

Participation in this study is complete after participant answers the final questionnaires.

Overall, this study should take about 30 minutes to complete.

This is an investigational study.

Up to 108 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced cancer diagnosis (locally advanced, recurrent or metastatic disease).
2. Patients presenting as follow-ups only at the outpatient Supportive Care Center.
3. Age >/= 18 years-old
4. English speaking

Exclusion Criteria:

1. Altered cognition (as assessed routinely in the Supportive Care Clinic using the Memorial Delirium Assessment Scale (MDAS), with a score of >/= 7/30).
2. Patients suffering from a severe psychiatric disorder or condition that would significantly interfere with study participation.
3. Patients with hearing and/or visual impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Participant's Perception of Physician's Compassion | 1 day
  Participant's rating of physician's compassion assessed by using a validated 5-item tool consisting of five 0-10 numerical rating scales assessing five dimensions: warm-cold, pleasant-unpleasant, compassionate- distant, sensitive- insensitive, and caring-uncaring.
  The sum of the five scales gives a final score representing physician's compassion on a scale of 0 to 50.

SECONDARY OUTCOMES:
Participant's Perception of Physician's Professionalism | 1 day
  Participant's rating of physician's professionalism assessed by using a validated 4-item tool assessing politeness, listening, explaining the condition and treatment to the patient and patient's involvement in treatment decisions. Participant rates from poor-1 to very good-5.
  The sum of these 4 items gives a final score representing physician's level of professionalism on a scale of 4 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Azhar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org